CLINICAL TRIAL: NCT07146165
Title: Clinical Evaluation of a New Platform for Bi-manual Endoscopic Resection in the Rectum and Sigma (EndoTEM)
Acronym: EndoTEM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Collaborators: Ovesco Endoscopy AG (Industry); Tuebingen Scientific Medical GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: S00830
Record Dates: First submitted 2025-07-31; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Adenoma Colon Polyp; Adenoma Colon
Keywords: endoscopic submucosal dissection; endoscopic en bloc resection; EndoTEM system; endoscopic portsystem; ESD
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoTEM-System (Experimental): Utilization of the EndoTEM system in the performance of routine endoscopic en bloc resection using endoscopic submucosal dissection.
  Interventions: Device: EndoTEM resection platform and technique

INTERVENTIONS:
Device: EndoTEM resection platform and technique — EndoTEM is a flexible transanally introduced port system that allows the insertion of a second instrument alongside the flexible endoscope. A curved rigid grasping instrument has been developed, with a 2 cm long tip that can be rotated and angled in all directions.
  Other Names: endoscopic portsystem

SUMMARY:
The goal of this clinical trial is to determine whether the use of the EndoTEM system during the endoscopic removal of polyps in the distal colon is feasible and safe.

The main questions it aims to answer are:

* Is the use of the EndoTEM system during the endoscopic removal of polyps in the distal colon feasible (i.e., does it enable complete resection of the polyp)?
* Is the use of the EndoTEM system during the endoscopic removal of polyps in the distal colon safe?

Participants will:

* be treated with the EndoTEM system during the endoscopic submucosal dissection of polyps in the distal colon.
* answere questionnaires on fecal continence and quality of life before and after the intervention.
* be treated following standard clinical procedures before, during and after the endoscopic removal.

ELIGIBILITY:
Inclusion Criteria:

* Availability of written informed consent from the patient
* Age > 18 years
* Adenoma or early carcinoma > 2 cm in the rectum or distal sigmoid colon with indication for endoscopic en bloc resection using endoscopic submucosal dissection

Exclusion Criteria:

* Informed consent not possible (e.g., language barrier)
* Stenoses or fistulas in the anal region
* Distance to the anocutaneous line ≤ 2 cm
* Distance to the anocutaneous line > 20 cm
* Individual medical assessment required for patients taking anticoagulant medication, in accordance with current ESGE guidelines
* Pregnancy or breastfeeding
* Vulnerable individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Technical success of the endoscopic resection | From the endoscopic resection to the follow-up endoscopy after 6 months.
  Macroscopically complete resection.

SECONDARY OUTCOMES:
R0 resection rate | Assessed with a biopsy collected during the intervention.
  Histological complete resection.
En bloc resection rate | Assessed during the intervention.
  Endoscopic removal of the polyp in one intact piece, including any necessary surrounding tissue.
Duration of the procedure | From endoscope insertion until the end of procedure including supplementary and prophylactic interventions.
Resection time | From start of the resection until detachment of the specimen.
Resection speed | Assessed during the intervention.
  Resected area per minute (mm²/min).
Periprocedural complications | Complications that occur during or immediately around the intervention (until 3-6 months post-intervention).
Requirement for surgical intervention | During the endoscopic submucosal dissection.
Rate of recurrence | Assessed during follow-up endoscopy 3-6 months post-intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Schmidt, Prof. Dr. med., Principal Investigator — Robert Bosch Krankenhaus GmbH
Locations (3):
- Germany (3):
  - Universitätsklinikum Freiburg, Klinik für Innere Medizin II, Freiburg im Breisgau
  - RKH Klinikum Ludwigsburg, Ludwigsburg
  - Robert Bosch Krankenhaus GmbH, Stuttgart

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueller J, Miedtke V, Kuellmer A et al. A novel endoscopic technique and device for bimanual rectosigmoidal ESD. Endoscopy 2023; 55(S02): 264 - 264. doi:10.1055/s-0043-1765725